CLINICAL TRIAL: NCT02638350
Title: Performance Evaluation of Clinical Ultrasound in Management of Acute Pulmonary Edema in Elderly Patient Over 65 Years, Admitted to a Host of Vital Emergency Services
Brief Title: Performance Evaluation of Clinical Ultrasound in Management of Acute Pulmonary Edema in Elderly Patient
Acronym: ECHOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/14/7423
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Edema; Respiratory Distress Syndrome
Keywords: lung ultrasound; Pulmonary Edema; Respiratory Distress Syndrome
MeSH Terms: conditions — Pulmonary Edema; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention lung ultrasound (Experimental): All patients will have strategy with lung ultrasoundlung ultrasound
  Interventions: Device: Strategy with lung ultrasound

INTERVENTIONS:
Device: Strategy with lung ultrasound — Each patient admitted for suspicion of acute lung edema will be treated according to the protocol of the emergency department.
  Another doctor will independently do a lung ultrasound and measurement of the inferior vena cava. The ultrasound results are not made available to the doctor in charge of the patient.
  At the end of the study, all the files will be analyzed by a independent committee, blinded ultrasound results for the final diagnosis of acute pulmonary edema.

SUMMARY:
The main objective is to assess the validation of the diagnosis early acute pulmonary edema in elderly patients with acute respiratory distress, admitted in a host of vital emergency services by lung ultrasound associated with the measurement of the inferior vena cava.

ELIGIBILITY:
Inclusion Criteria:

* Patient with compatible episode with acute edema (tachypnea with respiratory rate> 25/min and/or oxygen saturation on room air <90%, auscultation, dyspnea, sudden onset of symptoms)

Exclusion Criteria:

* Vital signs of distress requiring intubation tracheal immediately
* Myocardial infarction lower seat with extension to the right ventricle, in the acute phase

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
The result of lung ultrasound associated with the measurement of the inferior vena cava. | 2 hours
  Confirm the diagnosis of acute pulmonary edema associated with lung ultrasound to measure the inferior vena cava in patients aged over 65 years in acute respiratory distress, admitted to a service life-threatening emergencies.
  By checking the results of the ultrasound done by a different doctor from the one who took care of the patient.

SECONDARY OUTCOMES:
Number of the proportion of appropriate and inappropriate treatment. | 2 hours
  Comparison of specific treatments begun to emergency, as defined by the latest recommendations of Cardiology and Pneumology companies compared to the treatment that would have been given over the results of pulmonary ultrasound.
The duration of the medical care. | 2 hours
  The time between the patient support and the final diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Le Gourrierec, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, Midi Pyrenees, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zannad F, Mebazaa A, Juilliere Y, Cohen-Solal A, Guize L, Alla F, Rouge P, Blin P, Barlet MH, Paolozzi L, Vincent C, Desnos M, Samii K; EFICA Investigators. Clinical profile, contemporary management and one-year mortality in patients with severe acute heart failure syndromes: The EFICA study. Eur J Heart Fail. 2006 Nov;8(7):697-705. doi: 10.1016/j.ejheart.2006.01.001. Epub 2006 Mar 3. PMID 16516552
- [Background] Melniker LA, Leibner E, McKenney MG, Lopez P, Briggs WM, Mancuso CA. Randomized controlled clinical trial of point-of-care, limited ultrasonography for trauma in the emergency department: the first sonography outcomes assessment program trial. Ann Emerg Med. 2006 Sep;48(3):227-35. doi: 10.1016/j.annemergmed.2006.01.008. Epub 2006 Mar 24. PMID 16934640
- [Background] Nielsen LS, Svanegaard J, Wiggers P, Egeblad H. The yield of a diagnostic hospital dyspnoea clinic for the primary health care section. J Intern Med. 2001 Nov;250(5):422-8. doi: 10.1046/j.1365-2796.2001.00901.x. PMID 11887977
- [Background] Ray P, Birolleau S, Lefort Y, Becquemin MH, Beigelman C, Isnard R, Teixeira A, Arthaud M, Riou B, Boddaert J. Acute respiratory failure in the elderly: etiology, emergency diagnosis and prognosis. Crit Care. 2006;10(3):R82. doi: 10.1186/cc4926. Epub 2006 May 24. PMID 16723034
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136